CLINICAL TRIAL: NCT03078426
Title: LUNG MRI in the Management of Idiopathic Pulmonary Fibrosis : PIC'IRM
Brief Title: Lung MRI in the Management of Idiopathic Pulmonary Fibrosis
Acronym: PIC'IRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX2015/31
Record Dates: First submitted 2017-02-08; First posted 2017-03-13 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Lung; MRI; CT; Usual interstitial pneumonia; Ultra-short echo time
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Reference Standards

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 : UIP pattern (Experimental): 18 patients with UIP pattern at HRCT and IPF as a definite diagnosis.
  Interventions: Device: MRI; Other: Thoracic HRCT (standard reference)
- Group 2 : possible UIP pattern (Experimental): 7 patients with " possible " UIP pattern at HRCT with histopathology given by surgical lung biopsy making the diagnosis of IPF.
  Interventions: Device: MRI; Other: Thoracic HRCT (standard reference)
- Group 3 : diagnosis of fibrosing sarcoidosis (Experimental): 15 patients with the diagnosis of fibrosing sarcoidosis after multidisciplinary discussion.
  Interventions: Device: MRI; Other: Thoracic HRCT (standard reference)
- Group 4 : lung diseases without reticulations (Experimental): 20 patients with lung diseases without reticulations (acute or sub-acute hypersensitivity pneumonitis, organizing pneumonia, isolated pleural plaques) .
  Interventions: Device: MRI; Other: Thoracic HRCT (standard reference)

INTERVENTIONS:
Device: MRI — It will be performed on a 1.5-Tesla MR scanner (MAGNETOM Avanto, Siemens Healthcare, Erlangen, Germany). Acquisitions will be obtained in the axial plane using a 12-channel thorax/spine coil. Investigators will use previously published sequence parameters for each MRI sequence. PETRA will be acquired under free-breathing with respiratory gating at functional respiratory capacity.
Other: Thoracic HRCT (standard reference) — It will be performed on a 16 (Sensation 16, Siemens®) or 64 channels (Definition 64, Siemens®), without contrast agent injection.

SUMMARY:
High resolution computed tomography (HRCT) plays a major role in the management of idiopathic pulmonary fibrosis (IPF) by identifying characteristic lesions of usual interstitial pneumonia (UIP). Though HRCT is the standard reference to describe pulmonary structural alterations using a non invasive technique, it is nonetheless a radiating exam which provides limited functional information regarding inflammation. In this trial, the investigators aimed to evaluate whether MRI (Magnetic Resonance Imaging) using ultra-short echotime could be an alternative to HRCT in the assessment of the four morphological criteria required to define an UIP pattern. The investigators also planned to study the clinical value of the additional informations derived from MRI such as contrasts and lung perfusion using functional MRI.

DETAILED DESCRIPTION:
High resolution computed tomography (HRCT) is an essential component in the diagnostic pathway of idiopathic pulmonary fibrosis (IPF). With the appropriate clinical setting, the presence of an usual interstitial pneumonia (UIP) pattern on HRCT is sufficient to diagnose IPF. Four morphological criteria are required: (1) Subpleural, basal predominance, (2) Reticular abnormality, (3) Honeycombing with or without traction bronchiectasis, (4) Absence of features inconsistent with UIP pattern. However, HRCT is a radiating technique and only give data about structural alterations. Recent advances in three-dimensional ultra-short echo time (3D-UTE) imaging have shown promising results in improving lung MR (Magnetic Resonance) imaging quality. Since HRCT is the standard reference in IPF, the investigators aimed to evaluate whether thoracic MRI could be an alternative to HRCT in the assessment of the four radiologic criteria required for the diagnosis of IPF. Moreover, thoracic MRI could give new functional data, expected to relate to lung inflammation.

In order to study the diagnostic's accuracy of MRI for each radiological criteria defining UIP pattern, the investigators will compare HRCT and thoracic MRI of patients with IPF to HRCT and thoracic MRI of patients with other lung diseases that do not have all the UIP criteria.

Study procedure will be gadolinium-enhanced PETRA (pointwise encoding time reduction with radial acquisition) MR sequencing compared to unenhanced HRCT within 15 days. No follow-up is needed.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old followed in Bordeaux University Hospital
* Patients with a definite diagnosis of IPF :

  * Based on a "certain" UIP pattern at HRCT without histopathology
  * Based on a "possible" UIP pattern at HRCT with histopathology given by surgical lung biopsy.
* Patients with a diagnosis of fibrosing sarcoidosis after multidisciplinary discussion
* Patients with a diagnosis of acute or sub-acute hypersensitivity pneumonitis after multidisciplinary discussion
* Patients diagnosed with organizing pneumonia after multidisciplinary discussion
* Patients with a diagnosis of isolated pleural plaques after multidisciplinary discussion
* Patient able to withstand supine position for more than 30 minutes
* Patient affiliated to a social security system
* Patients who gave their written informed consent

Exclusion Criteria:

* Subject detained by judicial or administrative decision.
* Major protected by law.
* Subject not affiliated to a social security care
* Subject in period of relative exclusion in relation to another protocol.
* Patients with specific contraindication to undergoing MRI: iron material, a heart pacemaker, claustrophobia, gadolinium hypersensitivity, renal impairment with glomerular filtration rate less than 30 mL/min, pregnant or nursing woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
Measure of the diagnostic's accuracy of lung MRI compared to thoracic HRCT | Day 0
  Identifying the four radiologic criteria defining UIP pattern at inclusion (D0): (1) Subpleural, basal predominance, (2) Reticular abnormality, (3) Honeycombing with or without traction bronchiectasis, (4) Absence of features inconsistent with UIP pattern.

SECONDARY OUTCOMES:
Presence of the four radiologic criteria defining UIP pattern in the group of patient with definite diagnosis of IPF but with "possible" UIP pattern. | Day 0
Correlation between perfusion defects in MRI and IPF severity assessed by pulmonary function test : Forced Vital Capacity (FVC) | Day 0
Correlation between perfusion defects in MRI and IPF severity assessed by pulmonary function test : Transfer factor of carbon monoxide (TLCO) | Day 0
Correlation between perfusion defects in MRI and IPF severity assessed by 6 minutes exercise test | Day 0
Correlation between T2 signal intensity and IPF severity assessed by pulmonary function test : Forced Vital Capacity (FVC) | Day 0
Correlation between T2 signal intensity and IPF severity assessed by pulmonary function test : Transfer factor of carbon monoxide (TLCO) | Day 0
Correlation between T2 signal intensity and IPF severity assessed by 6 minutes exercise test | Day 0
Correlation between gadolinium-enhanced signal and IPF severity assessed by pulmonary function test : Forced Vital Capacity (FVC) | Day 0
Correlation between gadolinium-enhanced signal and IPF severity assessed by pulmonary function test : Transfer factor of carbon monoxide (TLCO) | Day 0
Correlation between gadolinium-enhanced signal and IPF severity assessed by 6 minutes exercise test | Day 0
The interobserver agreement of the results of the MRI will be estimated by the Kappa coefficient | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Elodie BLANCHARD, MD, Principal Investigator — University Hospital, Bordeaux; Rodolphe THIEBAUT, MD PhD, Study Chair — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Pessac, France

IPD SHARING:
Plan to Share IPD: No